CLINICAL TRIAL: NCT04307004
Title: Evaluating Novel Approaches for Estimating Awake and Sleep Blood Pressure - Better BP Study
Brief Title: Evaluating Novel Approaches for Estimating Awake and Sleep Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Columbia University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Emily B. Levitan, Professor and Vice Chair, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 5R01HL139716-02 (NIH); R01HL139716 (NIH)
Record Dates: First submitted 2020-03-02; First posted 2020-03-13 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Blood Pressure
Keywords: Ambulatory blood pressure monitoring; Home blood pressure monitoring; Clinic blood pressure; Blood pressure phenotypes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unattended vs Attended Blood Pressure (Other): Participants blood pressure will be measured three times attended and three times unattended using the Microlife WatchBP Office AFIB device. Whether investigators measure blood pressure attended first and then unattended or unattended first and then attended will be assigned using a random number generator. At visit 2, clinic blood pressure will be measured three times attended and three times unattended using the Microlife WatchBP Office AFIB device, as at visit 1, but in the reverse order.
  Interventions: Other: Unattended blood pressure measurement; Other: Attended blood pressure measurement
- ABPM vs HBPM (Other): Participants will be fitted with either the Microlife WatchBP O3 ambulatory blood pressure monitoring device or instructed on how to use the Microlife WatchBP Home N home blood pressure device, depending on which they are assigned to complete first. The order in which participants undergo ambulatory or home blood pressure monitoring will be assigned through a random number generator.
  Interventions: Other: Ambulatory blood pressure monitoring; Other: Home blood pressure monitoring

INTERVENTIONS:
Other: Unattended blood pressure measurement — Participants will have their blood pressure measured three times with an automated blood pressure monitor with a technician not present in the room.
  Other Names: Microlife WatchBP Office AFIB
  Arms: Unattended vs Attended Blood Pressure
Other: Attended blood pressure measurement — Participants will have their blood pressure measured three times with an automated blood pressure monitor with a technician present in the room.
  Other Names: Microlife WatchBP Office AFIB
  Arms: Unattended vs Attended Blood Pressure
Other: Ambulatory blood pressure monitoring — Participants will have their blood pressure measured every 30 minutes over 24-hours using an ambulatory blood pressure monitor.
  Other Names: Microlife WatchBP O3
  Arms: ABPM vs HBPM
Other: Home blood pressure monitoring — Participants will have their blood pressure measured three times overnight while they are asleep using a home blood pressure monitor.
  Other Names: Microlife WatchBP Home N
  Arms: ABPM vs HBPM

SUMMARY:
The purpose of the proposed study is to test whether measuring unattended blood pressure using an automated blood pressure monitor in a clinic setting without staff being present can reduce the need for assessing out-of- clinic awake blood pressure using ambulatory monitoring. Also, the investigators will test whether asleep blood pressure can be accurately measured using a novel home blood pressure monitoring device with less burden compared with ambulatory monitoring.

DETAILED DESCRIPTION:
For many people, blood pressure levels differ when measured in a doctor's office versus during normal daily activities. Ambulatory blood pressure monitoring, also called ABPM, involves wearing a blood pressure cuff attached to a device that is programmed to measure participants blood pressure every 30 minutes for a 24-hour period. ABPM can help better estimate a person's true average blood pressure. Although ABPM is recommended for diagnosing high blood pressure and it also measures blood pressure while people sleep, it is not available in many clinics and some people find the procedure to be uncomfortable. The purpose of this research study is to test whether blood pressure measured in a clinic setting without medical staff present is comparable to blood pressure levels measured during the daytime measured using an ABPM device. Also, the investigators will test whether asleep blood pressure can be accurately measured using a home blood pressure monitoring device. These findings may help identify new approaches for diagnosing high blood pressure without the need for ABPM. Each participant will complete four study visits. During the course of the study, participants will:

* Have their blood pressure measured in the clinic, six times at each of the first two study visits for a total of twelve blood pressure measurements.
* Complete questionnaires about their demographics, medical history, and participant sleeping habits.
* Have their blood drawn and provide a urine sample.
* Wear a Food and Drug Administration-approved ABPM device (Microlife WatchBP O3) for 24 hours.
* Wear a Food and Drug Administration-approved home blood pressure monitor (Microlife WatchBP Home N) while they sleep for one night.
* Wear an activity monitor (Actiwatch) for two 24-hour periods. The Actiwatch activity monitor measures activity levels and can be used to identify when they are asleep.
* Answer some questions about their experience while wearing the ABPM and home blood pressure monitor.
* Have an echocardiogram performed.

ELIGIBILITY:
Inclusion Criteria:

* Mean screening systolic blood pressure of 110 to < 160 mm Hg at most recent visit
* Mean screening diastolic blood pressure of 70 to <100 mm Hg at most recent visit

Exclusion Criteria:

* Currently taking antihypertensive medications
* Known to be currently pregnant
* History of sleep apnea
* History of heart attack, stroke, or any cardiovascular disease
* History of arrhythmia (e.g. - atrial fibrillation or ventricular tachycardia)
* Completed ambulatory blood pressure monitoring in the past year
* Second shift, overnight, or jobs that will not allow ambulatory blood pressure device to measure every 30 minutes for 24 hours.

Ages: 19 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Muntner, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham Hypertension Research Clinic, Birmingham, Alabama
  - Columbia University Medical Center - Hypertension Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cepeda M, Hubbard D, Oparil S, Schwartz JE, Jaeger BC, Hardy ST, Medina J, Chen L, Muntner P, Shimbo D. Evaluating novel approaches for estimating awake and sleep blood pressure: design of the Better BP Study - a randomised, crossover trial. BMJ Open. 2022 Jun 6;12(6):e058140. doi: 10.1136/bmjopen-2021-058140. PMID 35667722

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants whose systolic and diastolic blood pressure were 110 mm Hg to < 160 mm Hg and 70 mm Hg to <100 mm Hg, respectively, during screening. Participants were enrolled from a hypertension research clinic at the University of Alabama at Birmingham and a hypertension center at the Columbia University Medical Center. The first participant was enrolled on 7/15/2019 and the last participant was enrolled in 11/28/2022.
Pre-assignment Details: Of the 1,095 participants screened, 654 met the inclusion criteria and were randomized to either attended (technician present) before unattended (technician absent) blood pressure measurements or unattended before attended blood pressure measurements. The 654 participants were also randomized to undergo either Ambulatory Blood Pressure Monitoring before Home Blood Pressure Monitoring or Home Blood Pressure Monitoring before Ambulatory Blood Pressure Monitoring.
Groups:
- Attended Before Unattended BP: During visit 1, participants' clinic blood pressure was measured three times attended (i.e., in the presence of a technician) and then three times unattended (i.e., in the absence of a technician) using the Microlife WatchBP Office AFIB device. At visit 2, clinic blood pressure was measured three times unattended and then three times attended.
- Unattended Before Attended BP: During visit 1, participants' clinic blood pressure was measured three times unattended (i.e., in the absence of a technician) and then three times attended (i.e., in the presence of a technician) using the Microlife WatchBP Office AFIB device. At visit 2, clinic blood pressure was measured three times attended and then three times unattended.
- Ambulatory Blood Pressure Monitoring (ABPM) Before Home Blood Pressure Monitoring (HBPM): During visit 2, participants underwent 24 hours of Ambulatory Blood Pressure Monitoring (Microlife WatchBP O3) before undergoing one night of Home Blood Pressure Monitoring (Microlife WatchBP Home N) in visit 3.
- Home Blood Pressure Monitoring (HBPM) Before Ambulatory Blood Pressure Monitoring (ABPM): During visit 2, participants underwent one night of Home Blood Pressure Monitoring (Microlife WatchBP Home N) before undergoing 24 hours of Ambulatory Blood Pressure Monitoring (Microlife WatchBP O3) in visit 3.
Period: Randomization 1
Arm/Group | Attended Before Unattended BP | Unattended Before Attended BP | Ambulatory Blood Pressure Monitoring (ABPM) Before Home Blood Pressure Monitoring (HBPM) | Home Blood Pressure Monitoring (HBPM) Before Ambulatory Blood Pressure Monitoring (ABPM)
Started | 326 | 328 | 0 | 0
Completed | 301 | 302 | 0 | 0
Not Completed | 25 | 26 | 0 | 0
Not completed — Withdrawal by Subject | 25 | 26 | 0 | 0
Period: Randomization 2
Arm/Group | Attended Before Unattended BP | Unattended Before Attended BP | Ambulatory Blood Pressure Monitoring (ABPM) Before Home Blood Pressure Monitoring (HBPM) | Home Blood Pressure Monitoring (HBPM) Before Ambulatory Blood Pressure Monitoring (ABPM)
Started | 0 | 0 | 330 | 324
Completed | 0 | 0 | 302 | 301
Not Completed | 0 | 0 | 28 | 23
Not completed — Withdrawal by Subject | 0 | 0 | 28 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attended Before Unattended BP | Unattended Before Attended BP | Total
Number analyzed (Participants) | 301 | 302 | 603
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (16.0) | 37.9 (14.1) | 38.6 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 192 | 382
  Male | 111 | 110 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 29 | 69
  Not Hispanic or Latino | 259 | 272 | 531
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 39 | 51 | 90
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 64 | 68 | 132
  White | 150 | 141 | 291
  More than one race | 15 | 21 | 36
  Unknown or Not Reported | 33 | 20 | 53
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 301 | 302 | 603
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.8 (5.9) | 27.5 (5.8) | 27.2 (5.9)
Self-reported Hypertension [Count of Participants; unit: Participants] | 25 | 15 | 40
Sel-reported High Cholesterol [Count of Participants; unit: Participants] | 28 | 28 | 56
Sef-reported Diabetes [Count of Participants; unit: Participants] | 2 | 8 | 10
Self-reported Asthma or Hey Fever [Count of Participants; unit: Participants] | 32 | 36 | 68

OUTCOME MEASURES:

1. Primary Outcome: Absolute Difference Between Unattended and Attended Blood Pressure
Description: The difference between both systolic and diastolic blood pressure measurements when a technician is present versus when they are not present in the room.
Time Frame: 2 days
Population: Participants with complete attended and unattended blood pressure data.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Attended Clinic Systolic Blood Pressure: Systolic blood pressure collected by a clinic technician.
- Attended Clinic Diastolic Blood Pressure: Diastolic blood pressure collected by a clinic technician.
- Unattended Clinic Systolic Blood Pressure: Systolic blood pressure collected automatically in the clinic without a technician present.
- Unattended Clinic Diastolic Blood Pressure: Diastolic blood pressure collected automatically in the clinic without a technician present.
Arm/Group | Attended Clinic Systolic Blood Pressure | Attended Clinic Diastolic Blood Pressure | Unattended Clinic Systolic Blood Pressure | Unattended Clinic Diastolic Blood Pressure
Number analyzed (Participants) | 603 | 603 | 603 | 603
mm Hg | 119.5 (12.1) | 72.7 (7.8) | 118.7 (11.8) | 72.2 (7.7)
Statistical Analysis 1: Comparison: Attended Clinic Systolic Blood Pressure vs Unattended Clinic Systolic Blood Pressure; Test type: Superiority — The threshold for statistical significance was p = 0.05; p < 0.0001, Paired T Test, 2-sided; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [0.5 to 1.1] — Mean difference in systolic blood pressure = mean systolic blood pressure when attended - mean systolic blood pressure when not attended (i.e., unattended)
Statistical Analysis 2: Comparison: Attended Clinic Diastolic Blood Pressure vs Unattended Clinic Diastolic Blood Pressure; Test type: Superiority; p < 0.0001, Paired T Test, 2-sided — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.3 to 0.7] — Mean difference in diastolic blood pressure = mean diastolic blood pressure when attended - mean diastolic blood pressure when not attended (i.e., unattended)

2. Primary Outcome: Accuracy of Measuring Asleep Blood Pressure Using a Home Blood Pressure Monitor as Compared to Using an Ambulatory Blood Pressure Monitor
Description: Participants will have their systolic and diastolic blood pressure measured overnight using a home blood pressure monitor and over 24-hours using an ambulatory blood pressure monitor.
Time Frame: 2 days
Population: Participants with complete ambulatory and home blood pressure monitoring data.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Asleep Systolic Blood Pressure on Ambulatory Blood Pressure Monitoring: Asleep systolic blood pressure collected with an ambulatory blood pressure monitoring device.
- Asleep Diastolic Blood Pressure on Ambulatory Blood Pressure Monitoring: Asleep diastolic blood pressure collected with an ambulatory blood pressure monitoring device.
- Asleep Systolic Blood Pressure on Home Blood Pressure Monitoring: Asleep systolic blood pressure collected with a home blood pressure monitoring device.
- Asleep Diastolic Blood Pressure on Home Blood Pressure Monitoring: Asleep diastolic blood pressure collected with a home blood pressure monitoring device.
Arm/Group | Asleep Systolic Blood Pressure on Ambulatory Blood Pressure Monitoring | Asleep Diastolic Blood Pressure on Ambulatory Blood Pressure Monitoring | Asleep Systolic Blood Pressure on Home Blood Pressure Monitoring | Asleep Diastolic Blood Pressure on Home Blood Pressure Monitoring
Number analyzed (Participants) | 547 | 547 | 547 | 547
mm Hg | 104.1 (10.5) | 60.4 (7.5) | 106.4 (11.5) | 62.3 (8.3)
Statistical Analysis 1: Comparison: Asleep Systolic Blood Pressure on Ambulatory Blood Pressure Monitoring vs Asleep Systolic Blood Pressure on Home Blood Pressure Monitoring; Test type: Superiority; p < 0.0001, Paired T Test, 2-sided — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-3.0 to -1.5] — Mean difference in systolic blood pressure = mean systolic blood pressure on ambulatory blood pressure monitoring - mean systolic blood pressure on home blood pressure monitoring
Statistical Analysis 2: Comparison: Asleep Diastolic Blood Pressure on Ambulatory Blood Pressure Monitoring vs Asleep Diastolic Blood Pressure on Home Blood Pressure Monitoring; Test type: Superiority; p < 0.0001, Paired T Test, 2-sided — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.5 to -1.4] — Mean difference in diastolic blood pressure = mean diastolic blood pressure on ambulatory blood pressure monitoring - mean diastolic blood pressure on home blood pressure monitoring

3. Primary Outcome: Tolerability of Wearing a Home Blood Pressure Monitor Versus an Ambulatory Blood Pressure Monitor: Questionnaires
Description: Participants will complete questionnaires regarding their experience wearing both the ambulatory and home blood pressure monitors as well as a questionnaire on their willingness to wear the devices again.
Time Frame: 3 days
Population: Participants who completed questionnaires regarding their experiences wearing both the ambulatory and home blood pressure monitors.
Measure: Count of Participants; unit: Participants
Groups:
- Ambulatory Blood Pressure Monitoring: Experiences while undergoing ambulatory blood pressure monitoring
- Home Blood Pressure Monitoring: Experiences while undergoing home blood pressure monitoring
Arm/Group | Ambulatory Blood Pressure Monitoring | Home Blood Pressure Monitoring
Number analyzed (Participants) | 603 | 603
Participants
  Pain while wearing the monitor | 288 | 165
  Irritation while wearing the monitor | 410 | 258
  Bruising while wearing the monitor | 138 | 73
  Monitor was heavy to wear | 272 | 186
  Monitor was uncomfortable to wear | 508 | 467
  Monitor was straightforward to use | 590 | 584
  Monitor was cumbersome or awkward to wear | 507 | 404
  Noise of the monitor was disturbing to me | 193 | 173
  Noise of the monitor disturb others | 110 | 67
  Monitor was embarrassing to wear | 305 | 103
  Monitor interfered with normal sleeping pattern | 343 | 275
  Removed monitor due to disturbance while sleeping | 39 | 39

4. Secondary Outcome: Left Ventricular Mass Index
Description: Mean left ventricular mass index (LVMI)
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: g/m^2
Groups:
- Attended Before Unattended BP: Office blood pressure was measured by a clinic technician before automatically measured in the absence of a clinic technician
- Unattended Before Attended BP: Office blood pressure was automatically measured in the absence of a clinic technician before being measured by a clinic technician
- ABPM Before HBPM: Out-of-office blood pressure was measured on ABPM before being measured on HBPM
- HBPM Before ABPM: Out-of-office blood pressure was measured on HBPM before being measured on ABPM
Arm/Group | Attended Before Unattended BP | Unattended Before Attended BP | ABPM Before HBPM | HBPM Before ABPM
Number analyzed (Participants) | 301 | 302 | 302 | 301
g/m^2 | 67.6 (18.1) | 67.1 (16.9) | 66.9 (17.4) | 67.7 (17.5)
Statistical Analysis 1: Comparison: Attended Before Unattended BP vs Unattended Before Attended BP; We determined the association between attended systolic blood pressure and left ventricular mass index (LVMI). This analysis included 587 participants with attended office blood pressure measurements and valid LVMI measurements. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - Attended systolic blood pressure. Dependent variable - Left ventricular mass index; p < 0.001, Regression, Linear; beta coefficient = 0.43, 95% CI 2-sided [0.32 to 0.55], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Attended Before Unattended BP vs Unattended Before Attended BP; We determined the association between attended diastolic blood pressure measurements and left ventricular mass index (LVMI). This analysis included 587 with attended office blood pressure measurements and valid LVMI measurements. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - attended diastolic blood pressure. Dependent variable - left ventricular mass index; p < 0.001, Regression, Linear; beta coefficient = 0.42, 95% CI 2-sided [0.24 to 0.60], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Attended Before Unattended BP vs Unattended Before Attended BP; We determined the association between unattended systolic blood pressure and left ventricular mass index (LVMI). This analysis included 587 participants with unattended office blood pressure measurements and valid LVMI measurements. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - unattended systolic blood pressure. Dependent variable - left ventricular mass index; p < 0.001, Regression, Linear; beta coefficient = 0.44, 95% CI 2-sided [0.33 to 0.56], Standard Error of Mean 0.06
Statistical Analysis 4: Comparison: Attended Before Unattended BP vs Unattended Before Attended BP; We determined the association between unattended diastolic blood pressure and left ventricular mass index (LVMI). This analysis included 587 participants with unattended office blood pressure measurements and valid LVMI measurements. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - unattended diastolic blood pressure. Dependent variable - left ventricular mass index; p < 0.001, Regression, Linear; beta coefficient = 0.37, 95% CI 2-sided [0.19 to 0.55], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between awake systolic blood pressure from ambulatory blood pressure monitoring (ABPM) and left ventricular mass index (LVMI). This analysis included 554 participants with out-of-office blood pressure measurements and valid LVMI measurements. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - awake systolic blood pressure on ABPM Dependent variable - left ventricular mass index; p < 0.001, Regression, Linear; beta coefficient = 0.61, 95% CI 2-sided [0.47 to 0.74], Standard Error of Mean 0.07
Statistical Analysis 6: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between awake diastolic blood pressure on ambulatory blood pressure monitoring (ABPM) and left ventricular mass index (LVMI). This analysis included 554 participants with out-of-office blood pressure measurements and valid LVMI measurements. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - awake diastolic blood pressure on ABPM. Dependent variable - left ventricular mass index; p < 0.001, Regression, Linear; beta coefficient = 0.45, 95% CI 2-sided [0.25 to 0.66], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between asleep systolic blood pressure on home blood pressure monitoring (HBPM) and left ventricular mass index (LVMI). This analysis included 533 participants with HBPM data and valid LVMI. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - asleep systolic blood pressure on HBPM. Dependent variable - left ventricular mass index; p < 0.001, Regression, Linear; beta coefficient = 0.31, 95% CI 2-sided [0.19 to 0.44], Standard Error of Mean 0.06
Statistical Analysis 8: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between asleep diastolic blood pressure on home blood pressure monitoring (HBPM) and left ventricular mass index (LVMI). This analysis included 533 participants with data on HBPM and valid LVMI. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - asleep diastolic blood pressure on HBPM Dependent variable - left ventricular mass index; p = 0.01, Regression, Linear; beta coefficient = 0.23, 95% CI 2-sided [0.05 to 0.40], Standard Error of Mean 0.09
Statistical Analysis 9: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between asleep systolic blood pressure on ambulatory blood pressure monitoring (ABPM) and left ventricular mass index (LVMI). This analysis included 533 participants with data on ABPM and valid LVMI. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - asleep systolic blood pressure on ABPM. Dependent variable - left ventricular mass index; p < 0.001, Regression, Linear; beta coefficient = 0.45, 95% CI 2-sided [0.32 to 0.59], Standard Error of Mean 0.07
Statistical Analysis 10: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between asleep diastolic blood pressure on ambulatory blood pressure monitoring (ABPM) and left ventricular mass index (LVMI). This analysis included 533 participants with data on ABPM and valid LVMI. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - asleep diastolic blood pressure on ABPM Dependent variable - left ventricular mass index; p < 0.001, Regression, Linear; beta coefficient = 0.36, 95% CI 2-sided [0.16 to 0.55], Standard Error of Mean 0.10

5. Secondary Outcome: Urinary Albumin-to-creatine Ratio
Description: Mean urinary albumin-to-creatinine ratio (UACR)
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mg/g
Groups:
- Attended Before Unattended BP: Blood pressure was measured by a clinic technician before automatically measured in the absence of a clinic technician
- Unattended Before Attended BP: Blood pressure was measured automatically in the absence of a clinic technician before being measured by a clinic technician then urinary albumin and creatinine were collected and used to calculate urinary albumin-to-creatinine ratio.
Arm/Group | Attended Before Unattended BP | Unattended Before Attended BP | ABPM Before HBPM | HBPM Before ABPM
Number analyzed (Participants) | 301 | 302 | 302 | 301
mg/g | 21.7 (51.5) | 17.0 (21.6) | 19.7 (35.9) | 18.9 (43.0)
Statistical Analysis 1: Comparison: Attended Before Unattended BP vs Unattended Before Attended BP; We determined the association between attended systolic blood pressure and urinary albumin-to-creatinine ratio (UACR). This analysis included 555 participants with complete data on attended office blood pressure and UACR. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - attended systolic blood pressure. Dependent variable - urinary albumin-to-creatinine ratio; p = 0.17, Regression, Linear; beta coefficient = -0.20, 95% CI 2-sided [-0.47 to 0.08], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Attended Before Unattended BP vs Unattended Before Attended BP; We determined the association between attended diastolic blood pressure and urinary albumin-to-creatinine ratio (UACR). This analysis included 555 participants with complete data on attended office blood pressure and UACR. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - attended diastolic blood pressure. Dependent variable - urinary albumin-to-creatinine ratio; p = 0.20, Regression, Linear; beta coefficient = -0.28, 95% CI 2-sided [-0.70 to 0.15], Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Attended Before Unattended BP vs Unattended Before Attended BP; We determined the association between unattended systolic blood pressure and urinary albumin-to-creatinine ratio (UACR). This analysis included 555 participants with complete data on unattended blood pressure and UACR. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - unattended systolic blood pressure. Dependent variable - urinary albumin-to-creatinine ratio; p = 0.07, Regression, Linear; beta coefficient = -0.26, 95% CI 2-sided [-0.55 to 0.02], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Attended Before Unattended BP vs Unattended Before Attended BP; We determined the association between unattended diastolic blood pressure and urinary albumin-to-creatinine ratio (UACR). This analysis included 555 participants with complete data on unattended diastolic blood pressure and UACR. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - unattended diastolic blood pressure. Dependent variable - urinary albumin-to-creatinine ratio; p = 0.09, Regression, Linear; beta coefficient = -0.37, 95% CI 2-sided [-0.80 to 0.06], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between awake systolic blood pressure on ambulatory blood pressure monitoring (ABPM) and urinary albumin-to-creatinine ratio (UACR). This analysis included 523 participants with complete data on ABPM and UACR. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - awake systolic blood pressure on ambulatory blood pressure monitoring. Dependent variable - urinary albumin-to-creatinine ratio; p = 0.94, Regression, Linear; beta coefficient = 0.01, 95% CI 2-sided [-0.29 to 0.31], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between awake diastolic blood pressure on ambulatory blood pressure monitoring (ABPM) and urinary albumin-to-creatinine ratio (UACR). This analysis included 523 participants with complete data on ABPM and UACR. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - awake diastolic blood pressure on ambulatory blood pressure monitoring. Dependent variable - urinary albumin-to-creatinine ratio; p = 0.31, Regression, Linear; beta coefficient = 0.22, 95% CI 2-sided [-0.21 to 0.66], Standard Error of Mean 0.22
Statistical Analysis 7: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between asleep systolic blood pressure on home blood pressure monitoring (HBPM) and urinary albumin-to-creatinine ratio (UACR). This analysis included 505 participants with complete HBPM and UACR data. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - asleep systolic blood pressure on HBPM. Dependent variable - urinary albumin-to-creatinine ratio; p = 0.94, Regression, Linear; beta coefficient = -0.01, 95% CI 2-sided [-0.28 to 0.26], Standard Error of Mean 0.14
Statistical Analysis 8: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between asleep diastolic blood pressure on home blood pressure monitoring (HBPM) and urinary albumin-to-creatinine ratio (UACR). This analysis included 505 participants with complete HBPM and UACR data. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - asleep diastolic blood pressure on HBPM. Dependent variable - urinary albumin-to-creatinine ratio; p = 0.93, Regression, Linear; beta coefficient = -0.02, 95% CI 2-sided [-0.40 to 0.36], Standard Error of Mean 0.20
Statistical Analysis 9: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between asleep systolic blood pressure on ambulatory blood pressure monitoring (ABPM) and urinary albumin-to-creatinine ratio (UACR). This analysis included 505 participants with complete ABPM and UACR data. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - asleep systolic blood pressure on ABPM. Dependent variable - urinary albumin-to-creatinine ratio; p = 0.54, Regression, Linear; beta coefficient = 0.09, 95% CI 2-sided [-0.21 to 0.40], Standard Error of Mean 0.15
Statistical Analysis 10: Comparison: ABPM Before HBPM vs HBPM Before ABPM; We determined the association between asleep diastolic blood pressure on ambulatory blood pressure monitoring (ABPM) and urinary albumin-to-creatinine ratio (UACR). This analysis included 505 participants with complete ABPM and UACR data. This analysis combined across study arms as prespecified in the Study Protocol and Statistical Analysis Plan; Test type: Other — Independent variable - asleep diastolic blood pressure on ABPM. Dependent variable - urinary albumin-to-creatinine ratio; p = 0.23, Regression, Linear; beta coefficient = 0.26, 95% CI 2-sided [-0.16 to 0.68], Standard Error of Mean 0.21

ADVERSE EVENTS:
Time Frame: 2 weeks.
Arm/Group | Attended Before Unattended BP | Unattended Before Attended BP | Ambulatory Blood Pressure Monitoring (ABPM) Before Home Blood Pressure Monitoring (HBPM) | Home Blood Pressure Monitoring (HBPM) Before Ambulatory Blood Pressure Monitoring (ABPM)
All-Cause Mortality (participants affected / at risk) | 0/326 | 0/328 | 0/330 | 0/324
Serious Adverse Events (participants affected / at risk) | 0/326 | 0/328 | 0/330 | 0/324
Other Adverse Events (participants affected / at risk) | 0/326 | 0/328 | 228/330 | 244/324
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Attended Before Unattended BP (N=326) | Unattended Before Attended BP (N=328) | Ambulatory Blood Pressure Monitoring (ABPM) Before Home Blood Pressure Monitoring (HBPM) (N=330) | Home Blood Pressure Monitoring (HBPM) Before Ambulatory Blood Pressure Monitoring (ABPM) (N=324)
Brusing (Skin and subcutaneous tissue disorders) | 0 | 0 | 26 | 27
Pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 61 | 66
Irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 109 | 122
Discomfort (Skin and subcutaneous tissue disorders) | 0 | 0 | 190 | 208
Heavy to wear monitor (Skin and subcutaneous tissue disorders) | 0 | 0 | 73 | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT04307004/Prot_SAP_000.pdf